CLINICAL TRIAL: NCT05592704
Title: The Development and Application of a Toolset for Monitoring Personalized Physical Activity and Evaluation of Its Effectiveness in Individuals With Metabolic Syndrome
Brief Title: Remote Physical Activity Monitoring in Individuals With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PFAEV53
Record Dates: First submitted 2022-09-28; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-09

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Physical activity; Telemonitoring; Smartphone application; Wearables; Cardiovascular prevention; mHealth; Digital health
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Individuals participated in the 2-month outpatient aerobic exercise training program, which consisted of 40 training sessions on a cycle ergometer 5 times/week for 40 min. Then during motivational consultation, individuals received recommendations for healthy lifestyle and home-based training. After that, study subjects participated in the 6-month home-based aerobic exercise program using wearable device (heart rate monitor), which was connected to the smartphone via Bluetooth. A special smartphone application enabled participants to keep their training heart rate during home-based exercises (or workouts).
  Interventions: Device: Usage of a wearable heart rate monitor and a smartphone with the application for home-based exercises
- Control group (No Intervention): Individuals participated in the 2-month outpatient aerobic exercise training program, which consisted of 40 training sessions on a cycle ergometer 5 times/week for 40 min. Then during motivational consultation, individuals received recommendations for healthy lifestyle and home-based training. After that, study subjects participated in the 6-month home-based aerobic exercise program without wearable devices and smartphone application.

INTERVENTIONS:
Device: Usage of a wearable heart rate monitor and a smartphone with the application for home-based exercises — Physical activity self-monitoring using a wearable heart rate monitor and a smartphone with specially designed application
  Arms: Intervention group

SUMMARY:
A prospective intervention study to evaluate the effectiveness of the developed toolset for remote physical activity monitoring to improve arterial stiffness and other cardiometabolic parameters and to increase physical activity levels and the compliance to the prescribed exercise in individuals with metabolic syndrome.

DETAILED DESCRIPTION:
At first, all subjects of the prospective study participated in the 2-month outpatient aerobic exercise program, which consisted of 40 aerobic training sessions on a cycle ergometer 5 times/week for 40 min. During all training sessions, heart rate was maintained at the targeted level, which was obtained individually by cardiopulmonary test. After 2 months, during individual motivational consultations, all participants received recommendations for home-based training and were randomly allocated to the intervention or the control group. Then only the intervention group subjects participated in the 6-month home-based aerobic exercise program using a wearable heart rate monitor, which was connected to the smartphone via Bluetooth. The intervention group subjects used a smartphone application created for the study. The control group participants were asked to exercise at home for 6 months without wearables and smartphone application. The evaluation of the study participants was performed at baseline (1st visit), after 2 months (2nd visit) and after 8 months (3rd visit).

ELIGIBILITY:
Inclusion Criteria:

* Males (40-55 years) and females (50-65 years) with metabolic syndrome, having at least three of the following five criteria: hypertriglyceridemia (triglycerides ≥ 1.7 mmol/l); high-density lipoprotein cholesterol ≤ 1.03 mmol/l for men or ≤ 1.29 mmol/l for women; abdominal obesity (waist circumference > 102 cm for men and > 88 cm for women); elevated blood pressure (systolic blood pressure ≥ 130 mmHg and/or diastolic blood pressure ≥ 85 mmHg or current use of antihypertensive drugs); elevated fasting plasma glucose ≥ 5.6 mmol/l;

Exclusion Criteria:

* Patients with overt cardiovascular disease (previous myocardial infarction, coronary artery bypass surgery, percutaneous coronary intervention, previous stroke)
* Patients with severe heart failure symptoms, uncontrolled hypertension
* Patients with urinary tract infection or fever for another unknown reason
* Patients who have actively exercised in the last 24 hours
* Pregnant women

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in carotid-radial pulse wave velocity and carotid-femoral pulse wave velocity | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Measured by applanation tonometry (SphygmoCor, ArtCor Medical, Sydney, Australia), all in m/s.
Changes in mean blood pressure in the aorta, mean blood pressure in the brachial artery and pulse pressure in the aorta | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Measured by applanation tonometry (SphygmoCor, ArtCor Medical, Sydney, Australia), all in mmHg.
Changes in cardio-ankle vascular index | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Measured by VaSera-1000 (Fukuda, Denshi, Japan).
Changes in common carotid artery intima-media thickness | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Measured by performing a carotid artery ultrasound (in μm).
Changes in carotid artery ß stiffness index | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Measured by performing a carotid artery ultrasound.
Changes in maximal oxygen consumption (VO2max) | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Measured by performing a cardiopulmonary exercise test (Vmax® Encore 229, SensorMedics, USA) in ml/kg/min.
Changes in the levels of metabolic equivalents of task (METs) | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Measured by performing a cardiopulmonary exercise test (Vmax® Encore 229, SensorMedics, USA) in METs.
Changes in heart rate at rest and training heart rate | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Measured by performing a cardiopulmonary exercise test (Vmax® Encore 229, SensorMedics, USA) in bpm.
Changes in lipids and glucose levels in the blood | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Total cholesterol, triglycerides, low density lipoprotein-cholesterol, high density lipoprotein-cholesterol levels and fasting glucose were measured in blood samples (all in mmol/L).
Changes in C-reactive protein levels in the blood | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Measured in blood samples (in mg/L).
Changes in body mass index (BMI) | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Weight (kg) and height (m) were measured to report BMI in kg/m^2.
Changes in waist circumference | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Waist circumference was measured in cm.
Changes in blood pressure parameters | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Systolic and diastolic blood pressure (in mmHg) were measured in a sitting position using oscillometric device.
Changes in the status of cardiovascular risk factors | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Smoking status (smoking < 10 cigarettes/day (yes/no), smoking > 10 cigarettes/day (yes/no), non-smoking (yes/no), smoking cessation (yes/no)), arterial hypertension status (yes/no), dyslipidaemia status (yes/no) were assessed in medical records.
Changes in health-related quality of life | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  Health-related quality of life was evaluated by the Medical Outcomes Study 36-Item Short-Form Health Survey. In this questionnaire, each domain of health-related quality of life is scored from 0 to 100 (100 points show the best estimate).
Changes in motivation for physical activity | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  The motivation for physical activity was evaluated by the Exercise Motivations Inventory-2 (EMI-2). In this questionnaire, the answer to each statement is given on a six-step scale from 0 points ("not at all true for me") to 5 points ("very true for me"). Higher mean scores in the appropriate items of the 14 subscales indicate better result.
Changes in the levels of anxiety and depression | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  The levels of anxiety and depression were evaluated by the Hospital Anxiety and Depression scale, where 8-10 scores indicate mild, 11-14 scores - moderate, and 15-21 scores - severe anxiety or depression.
Changes in the levels of self-reported physical activity | After 2 months (between 1st and 2nd visit), after 6 months (between 2nd and 3rd visit), after 8 months (between 1st visit and 3rd visit)
  The levels of self-reported physical activity (in minutes/week) were measured by using the International Physical Activity Questionnaire short form (IPAQ-sf). Higher values indicate better result.

SECONDARY OUTCOMES:
Changes in the levels of objectively measured physical activity | After 6 months (between 2nd and 3rd visit)
  Total duration of physical activity (in minutes) and duration of physical activity divided by the type and timing of workout (in minutes) were measured by the real-time physical activity data received through the smartphone application.
Changes in the number of workouts | After 6 months (between 2nd and 3rd visit)
  Total number of workouts and number of workouts divided by the type and timing of workout were measured by the real-time physical activity data received through the smartphone application.
Changes of compliance to the prescribed exercise in terms of workout duration | After 6 months (between 2nd and 3rd visit)
  The average workout duration (in minutes) was measured by the real-time physical activity data received through the smartphone application. Higher values indicate better compliance.
Changes of compliance to the prescribed exercise in terms of intensity | After 6 months (between 2nd and 3rd visit)
  The proportion (%) of the workout time in prescribed exercise intensity was measured by the real-time physical activity data received through the smartphone application. Higher values indicate better compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandras Laucevicius, PhD, Principal Investigator — Clinic of Cardiac and Vascular Diseases, Faculty of Medicine, Vilnius University
Locations (1):
- Outpatient clinic "InMedica", Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zupkauskiene J, Lauceviciene I, Ryliskyte L, Navickas P, Kizlaitis R, Laucevicius A. Ambulatory and successive home-based heart rate targeted aerobic training improves arterial parameters: a follow-up study in people with metabolic syndrome. Ann Med. 2023;55(2):2250363. doi: 10.1080/07853890.2023.2250363. PMID 37625386